CLINICAL TRIAL: NCT03600922
Title: A Prospective Randomized Clinical Study of Patellar Resurfacing and Non-resurfacing in One-stage Bilateral Total Knee Arthroplasty
Brief Title: Clinical Study of Patellar Resurfacing and Non-resurfacing in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaocheng People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCHOSPITAL-123456
Record Dates: First submitted 2018-06-01; First posted 2018-07-26 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Total Knee Arthroplasty
Keywords: Osteoarthritis; Patellar resurfacing; Anterior knee pain
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental)
  Interventions: Procedure: the patella was resurfaced.

INTERVENTIONS:
Procedure: the patella was resurfaced. — Patellar resurfacing was undertaken using a cemented, inset domed component in TKA.

SUMMARY:
The literature regarding resurfacing of the patella in total knee arthroplasty has conflicting conclusions. This study assesses medium-term clinical results of total knee arthroplasties performed with and without the patellar resurfacing in patients undergoing single-staged bilateral total knee arthroplasty in a randomized controlled, clinical study at a minimum of 5 years follow-up.

DETAILED DESCRIPTION:
Sixty-six patients (132 knees) underwent primary single-staged bilateral total knee arthroplasty for osteoarthritis. Patients were randomized to receive resurfacing or retention of the patella. All patients received the Scorpio NRG knee prosthesis. Evaluations were done preoperatively and yearly, up to a minimum of 5 years postoperatively. Knee Society Score and Feller Score outcomes were measured. Anterior knee pain, the clunk of patella, and patient satisfaction questionnaires were completed.

ELIGIBILITY:
Inclusion Criteria:

* degenerative OA
* 50-75 years
* All patients with OA were bilateral knee OA

Exclusion Criteria:

* previous patellectomy
* inflammatory arthritis
* patellar fracture
* patellar instability
* previous extensor mechanism procedures
* high tibial osteotomy,
* severe valgus or varus deformity (> 20°), severe flexion contracture (> 30°)
* previous unicondylar knee replacement
* a history of septic arthritis or osteomyelitis.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in the Feller score | Baseline,1,2,3,4 and 5 years
  The Feller score consists four parts.Total score is 30 score (0-30) and the higher values represent a better outcome. The Feller score has points for Anterior knee pain (0 worst-15 best), quadriceps strength (1 worst -5 best) , ability to rise from chairand stability(0 worst-5 best )and stair-climbing(2 worst-5 best ). The scores from each item are summed to produce a total score
Change From Baseline in visual analogue scale (VAS) | Baseline,1,2,3,4 and 5 years
  The Visual analogue scale (VAS)is ranging from 0 to 10 points, with 0 being no pain and 10 being maximum pain.The higher values represent a worse outcome.
Change From Baseline in knee society score ( KSS) | Baseline,1,2,3,4 and 5 years
  The knee society score ( KSS) which consists of a 100-point scale for knee score and 100-point score for function score. The knee score has points for pain (0 worst -50 best ), range of motion (0 worst -25 best ) and stability (0 worst -25 best ). scores from each item are summed to produce a total score .The function score has points for walking ability (0 worst -50 best ) and stair climbing ability (0 worst -50 best ), scores from each item are summed to produce a total score.The knee score and the function score are recorded respectively.The higher values represent a better outcome.
Change From Baseline in anteroposterior long weight-bearing X-ray | Baseline,1,2,3,4 and 5 years
  anteroposterior long weight-bearing X-ray
Change From Baseline in MOS item short from health survey(SF-36) | Baseline,1,2,3,4 and 5 years
  The MOS item short from health survey(SF-36) was constructed to survey health status in the Medical Outcomes Study. The SF-36 was designed for use in clinical practice and research, health policy evaluations, and general population surveys. The SF-36 includes one multi-item scale that assesses eight health concepts: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions.

REFERENCES:
- [Derived] Ha C, Wang B, Li W, Sun K, Wang D, Li Q. Resurfacing versus not-resurfacing the patella in one-stage bilateral total knee arthroplasty: a prospective randomized clinical trial. Int Orthop. 2019 Nov;43(11):2519-2527. doi: 10.1007/s00264-019-04361-7. Epub 2019 Jun 21. PMID 31227852